CLINICAL TRIAL: NCT00840047
Title: Methionine PET/CT Studies In Patients With Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: METPET; NCI-2011-02414 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Brain Tumors and/or Solid Tumors Including; Brain Stem Glioma; High Grade CNS Tumors; Ependymoma; Medulloblastoma; Craniopharyngioma; Low Grade CNS Tumors; Hodgkin Lymphoma; Non Hodgkin Lymphoma; Ewing Sarcoma; Osteosarcoma; Rhabdomyosarcoma; Neuroblastoma; Other
Keywords: Pediatric brain tumor; Pediatric solid tumor; Pediatric solid neoplasms
MeSH Terms: conditions — Ependymoma; Medulloblastoma; Craniopharyngioma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Sarcoma, Ewing; Osteosarcoma; Rhabdomyosarcoma; Neuroblastoma | interventions — Methionine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Participants who meet the eligibility criteria in the study will receive methionine.
  Interventions: Drug: Methionine

INTERVENTIONS:
Drug: Methionine — Intravenous injection
  Other Names: MET; [11C]-L-Methionine

SUMMARY:
The purpose of this study is to test the usefulness of imaging with radiolabeled methionine in the evaluation of children and young adults with tumor(s). Methionine is a naturally occurring essential amino acid. It is crucial for the formation of proteins. When labeled with carbon-11 (C-11), a radioactive isotope of the naturally occurring carbon-12, the distribution of methionine can be determined noninvasively using a PET (positron emission tomography) camera. C-11 methionine (MET) has been shown valuable in the monitoring of a large number of neoplasms. Since C-11 has a short half life (20 minutes), MET must be produced in a facility very close to its intended use. Thus, it is not widely available and is produced only at select institutions with access to a cyclotron and PET chemistry facility. With the new availability of short lived tracers produced by its PET chemistry unit, St. Jude Children's Research Hospital (St. Jude) is one of only a few facilities with the capabilities and interests to evaluate the utility of PET scanning in the detection of tumors, evaluation of response to therapy, and distinction of residual tumor from scar tissue in patients who have completed therapy. The investigators propose to examine the biodistribution of MET in patients with malignant solid neoplasms, with emphasis on central nervous system (CNS) tumors and sarcomas. This project introduces a new diagnostic test for the noninvasive evaluation of neoplasms in pediatric oncology. Although not the primary purpose of this proposal, the investigators anticipate that MET studies will provide useful clinical information for the management of patients with malignant neoplasms.

DETAILED DESCRIPTION:
The study focuses on the following objectives:

Primary objective:

* To estimate the success rate of Methionine (MET) for visualizing tumors at the time of diagnosis. The study hypothesizes that at least 70% of newly diagnosed tumors within each group will be studied and will be successfully visualized.

Secondary objective:

* To compare uptake of MET in tumors with tumor grade in patients with newly diagnosed or relapsed, and/or persistent disease. Hypothesis: high grade tumors will concentrate higher amounts of MET than lower grade tumors measured both qualitatively and semi-quantitatively.
* To examine the bio-distribution of MET in organs that do not contain tumor, in particular the lungs, heart, mediastinum, liver, spleen, pancreas, muscle, brain, and bone marrow.

Exploratory objectives:

* To compare the findings on MET PET scans with those of standard imaging modalities, principally MRI (magnetic resonance imaging) and FDG (fluorodeoxyglucose) PET CT (computed tomography) at diagnosis, or at study enrollment for patients with relapsed and or persistent disease, and for all patients over time.
* To compare the extent of abnormality on MRI with that of MET.
* To determine the presence or absence of elevated MET uptake beyond those of MRI defined abnormality.
* To explore the relationship between MET uptake and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* All participants under the care of St. Jude physicians with known or suspected neoplastic disease are eligible for participation.
* Participants will have had, or are scheduled to have clinical imaging evaluations which may include FDG PET CT, or CT, or MRI within 4 weeks of entry.
* No limit on age or gender.
* Female participants of childbearing age must not be lactating due to theoretical potential harm to the infant from exposure to radiation.
* Informed consent signed by participant, parent, or guardian according to the guidelines of the institutional review board.

Exclusion Criteria:

* More than 6 MET PET scans within the previous 12 months.
* Inability or unwillingness of research participant, parent, or legal guardian/representative to give written informed consent.

Inclusion Criteria for Open-Access

* All participants under the care of St. Jude physicians with known or suspected neoplastic disease are eligible for participation.
* No limit on age or gender
* Female participants of childbearing age must not be lactating due to theoretical potential harm to the infant from exposure to radiation.
* Informed consent signed by participant, parent, or guardian according to the guidelines of the institutional review board.

Exclusion Criteria for Open-Access

* More than 6 MET PET scans within the previous 12 months.
* Inability or unwillingness of research participant, parent, or legal guardian/representative to give written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 503 (Actual)
Dates: Start 2009-07-20 (Actual); Primary Completion 2027-07-27 (Estimated); Study Completion 2027-07-27 (Estimated)

PRIMARY OUTCOMES:
Success rate of methionine (MET) for visualizing tumors | Baseline
  To estimate the success rate of methionine (MET) for visualizing tumors at the time of diagnosis. We hypothesize that at least 70% of tumors within each group studied will be successfully visualized.

SECONDARY OUTCOMES:
Association of methionine uptake with tumor grade | End of study (maximum of 3 years post methionine infusion and PET scan)
  Methionine uptake in tumors will be compared among tumor grades in patients with newly diagnosed or relapsed, and/or persistent disease. Hypothesis: high-grade tumors will concentrate higher amounts of MET than lower-grade tumors measured both qualitatively and semi-quantitatively.
Bio-distribution of MET in organs | At baseline, after enrollment of the first 93 participants
  Whole body scans will be acquired and descriptive statistics for MET uptake from other parts of the body will be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Barry L Shulkin, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

DOCUMENTS (1):
  • Informed Consent Form (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/47/NCT00840047/ICF_000.pdf